CLINICAL TRIAL: NCT07198867
Title: A Study of A-CAR028 Treatment in Subjects With Relapsed/ Refractory Acute Myeloid Leukemia
Brief Title: A Study of A-CAR028 Treatment in Subjects With Relapsed or Refractory Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Shanghai AbelZeta Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1207-047
Record Dates: First submitted 2025-07-30; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia (AML); CAR-T Cell Therapy
Keywords: A-CAR028; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A-CAR028 (Experimental): Autologous A-CAR028 administered by intravenous (IV) infusion
  Interventions: Biological: A-CAR028

INTERVENTIONS:
Biological: A-CAR028 — A-CAR028 is a novel 2nd generation 4-1BB bispecific chimeric antigen receptor T-cell (CAR-T) targeting both CD33 and CLL-1 antigens

SUMMARY:
This is a single-center, open-label study to evaluate the safety and efficacy of A-CAR028 in relapsed/refractory acute myeloid leukemia patients

DETAILED DESCRIPTION:
The study includes the following sequential phases: Screening, Apheresis and A-CAR028 manufacturing, Baseline testing, Lymphodepletion, A-CAR028 infusion, Dose-limiting toxicity observation and Follow-up Visit

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old at the time of signing the Informed Consent Form (ICF)
* More than 12 weeks of expected survival
* ECOG score 0 or 1
* Relapsed or refractory AML
* Adequate organ function

Exclusion Criteria:

* Acute Promyelocytic Leukemia (APL)
* Mixed Phenotype Acute Leukemia (MPAL)
* Acute Undifferentiated Leukemia (AUL)
* Only extramedullary leukemia
* Known allergies to the components or excipients of the A-CAR028 cell product
* Severe heart diseases, including but not limited to, myocardial infarction, angioplasty or stent implantation within 12 months prior to signing the ICF, unstable angina pectoris, severe arrhythmia, history of severe non-ischemic cardiomyopathy, heart failure
* Autologous or allogeneic hematopoietic stem cell transplantation within 3 months prior to signing the ICF
* Central nervous system (CNS) involvement or symptoms of CNS involvement (including cranial nerve lesions and extensive lesions or spinal cord compression)
* A stroke or seizure occurred within 12 months prior to signing the ICF
* Malignancy history within 5 years prior to signing the ICF
* Uncontrolled active infection
* Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV), Treponema Pallidum (TP) positive, Cytomegalovirus (CMV) DNA positive
* Live vaccine injection within 4 weeks prior to signing the ICF
* Acute or chronic graft-versus-host disease (GVHD) was present at screening
* Inadequate washing time for previous treatment
* Previously treated with CAR-T cell products or genetically modified T cell therapies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | Throughout the 28 days post A-CAR028 infusion
Incidence and severity of Treatment Emergent Adverse Events (TEAEs) | Throughout the 3 months post A-CAR028 infusion

SECONDARY OUTCOMES:
Incidence and severity of Adverse Events (AEs) | Throughout the 2 years post A-CAR028 infusion
Overall Response Rate (ORR): including Complete Response (CR), CR with Partial Hematologic Recovery (CRh), CR with Incomplete Hematologic Recovery (CRi), Morphologic Leukemia-free State (MLFS) and Partial Response (PR) | Throughout the 2 years post A-CAR028 infusion
Duration of Response (DOR) | Throughout the 2 years post A-CAR028 infusion
Event-free Survival (EFS) | Throughout the 2 years post A-CAR028 infusion
Overall Survival (OS) | Throughout the 2 years post A-CAR028 infusion
Maximal plasma concentration (Cmax) | Throughout the 2 years post A-CAR028 infusion
Time to reach the maximal plasma concentration (Tmax) | Throughout the 2 years post A-CAR028 infusion
Area under the curve within 28 days (AUC0-28d) | Throughout the 2 years post A-CAR028 infusion
Time of last measurable observed concentration (Tlast) | Throughout the 2 years post A-CAR028 infusion
Changes of CD33/CLL-1 positive cells in bone marrow | Throughout the 2 years post A-CAR028 infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology, The First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No